CLINICAL TRIAL: NCT06910150
Title: Immediate Effectiveness of a Single Session of Analgesic Electrostimulation on the Femoral Quadriceps in Patients After Anterior Cruciate Ligament Reconstruction: A Randomized Clinical Trial.
Brief Title: Effectiveness of a Session of Analgesic Electrostimulation (Invasive and Non-invasive) Applied to the Quadriceps Muscle in Patients After Knee Surgery.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Javier Reina Abellan; PhD, Principal Investigator at Universidad Católica San Antonio de Murcia, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE112417
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Long-Term Potentiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Participants will only undergo a conventional physiotherapy rehabilitation program for anterior cruciate ligament rehabilitation.
- Experimental Group 1 (Experimental): Participants will undergo a conventional anterior cruciate ligament rehabilitation physiotherapy program and receive a single session of analgesic transcutaneous electrical nerve stimulation (TENS).
  Interventions: Procedure: Non-invasive analgesic electrostimulation
- Experimental Group 2 (Experimental): Participants will undergo a conventional anterior cruciate ligament rehabilitation physiotherapy program and receive a single session of invasive analgesic electrostimulation (LTP, long-term potentiation).
  Interventions: Procedure: Invasive analgesic electrostimulation

INTERVENTIONS:
Procedure: Non-invasive analgesic electrostimulation — A single session of non-invasive analgesic electrostimulation is applied to the motor points of the vastus medialis and vastus lateralis muscles of the quadriceps femoris in patients who had undergone anterior cruciate ligament reconstruction. A biphasic, symmetrical, square-wave current is used at a frequency of 100 Hz, a pulse width of 200 μs, and an intensity adjusted to the patient's pain threshold, applied for 30 minutes.
  Other Names: TENS (Transcutaneous Electrical Nerve Stimulation)
  Arms: Experimental Group 1
Procedure: Invasive analgesic electrostimulation — A single session of invasive analgesic electrostimulation is applied to a motor point of the vastus medialis of the quadriceps femoris in patients who had undergone anterior cruciate ligament reconstruction. A biphasic, symmetrical, square-wave current is used at a frequency of 100 Hz, a pulse width of 250 μs, and an intensity defined as perceptible to the patient but never painful (200 μA above the detection threshold for each subject).
  Other Names: LTP protocol (long-term potentiation)
  Arms: Experimental Group 2

SUMMARY:
The anterior cruciate ligament (ACL) injury is one of the most prevalent injuries in the musculoskeletal system. Consequently, its surgical reconstruction is among the most commonly performed procedures in current clinical practice.

The aim of this clinical trial is to investigate if the application of a single session of electrical currents to the quadriceps muscle can reduce pain in individuals who have undergone ACL surgery. Additionally, the trial will assess whether this intervention increases the pressure pain threshold, mobility, strength and functionality of the operated knee, as well as improving the participant's quality of life. Effusion and edema of the operated knee will also be measured.

Participants in this clinical trial will be randomly assigned to three study groups: one control group and two experimental groups.

All participants will undergo a conventional physiotherapy program for knee rehabilitation. This program includes manual therapy with a physiotherapist and exercises aimed at strengthening the CORE, hip and knee muscles.

Participants in the first experimental group will receive an additional session of superficial (non-invasive) electrical currents applied to the quadriceps muscle of the operated knee.

Participants in the second experimental group will receive an additional session of invasive electrical currents applied to the quadriceps muscle of the operated knee.

Each patient will be assessed four times: before the intervention, immediately after the intervention, and 1 and 7 days post-intervention. Functionality of the operated knee and quality of life will only be assessed before the intervention and 7 days post-intervention using self-reported scales.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 55 years, regardless of gender.
* Subjects who have undergone surgical ACL reconstruction within the past six weeks, with or without additional procedures on one or both menisci due to their high concomitance, and with or without Lemaire reinforcement in the form of extra-articular lateral tenodesis.
* Subjects experiencing pain in the operated knee.
* Voluntary signing of the informed consent form for the study.

Exclusion Criteria:

* Contraindications for invasive therapies:
* Subjects with chronic joint pathology.
* Subjects with prostheses or osteosynthesis in the affected lower limb.
* Subjects with heart disease.
* Subjects with neoplasms.
* Subjects with coagulopathies.
* Subjects with epilepsy.
* Subjects with pacemakers.
* Pregnant patients.
* Subjects with belonephobia (severe fear of needles).
* Subjects with neuropathic pain.
* Subjects with central nervous system disorders.
* Subjects with a history of neurological disorders.
* Subjects with a history of lumbar hernia or protrusion due to a possible involvement of the lumbar plexus.
* Subjects with a history of spinal surgery.
* Subjects presenting any bilateral symptoms.
* Subjects with a BMI greater than 30 kg/m².
* Subjects taking analgesic medication.
* Subjects receiving any alternative treatment not proposed in this study, which could alter the results.
* Subjects scoring above 37.5 points on the "Personal Psychological Apprehension Scale in Physiotherapy".
* Contraindications for dynamometric measurement:
* Subjects with acute quadriceps muscle injury.
* Subjects with joint instability.
* Subjects with acute joint inflammation.
* Subjects who voluntarily withdraw from the study.
* Subjects absent for any measurement session.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in knee pain from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed with the Numeric Rating Scale (NRS). The patient reports their pain at the moment of measurement on a scale from 0 (no pain) to 10 (worst imaginable pain).
Change in knee range of movement from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed with a manual universal goniometer.
Change in knee pain threshold to pressure from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed with an analog algometer (FPK 20).
Change in maximum isometric quadriceps strength from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed with a portable handheld dynamometer Lafayette© (Lafayette Manual Muscle Tester, Lafayette Instruments, Lafayette, IN)
Change in thigh muscle atrophy from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed with a flexible measuring tape.
Change in knee intra-articular effusion from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed on the basis of bulge and dancing patella signs and reported as 3 (>60 cm3 - tight capsule), 2 (25-60 cm3 - visible), 1(<25 cm3 - palpable by smoothing out the joint capsule), or 0 (no effusion).
Change in knee extra-articular edema from baseline to immediately after the intervention, as well as at one and seven days post-intervention. | From baseline to immediately after the intervention, as well as at one and seven days post-intervention.
  Assessed with a flexible measuring tape.
Change in quality of life from baseline to seven days post-intervention. | From baseline to seven days post-intervention.
  Assessed with the self-reported scale "Anterior Cruciate Ligament - Quality of Life - Spanish".
  Potential score: 0-3200. The higher the score, the better the patient's quality of life..
Change in knee functionality from baseline to seven days post-intervention. | From baseline to seven days post-intervention.
  Assessed with the self-reported questionnaire "Lysholm Scale". Potential score: 0-100 points. The higher the score, the better the patient's functionality.
Needle apprehension at baseline | At baseline
  Assessed with the self-reported questionnaire "Personal Psychological Apprehension Scale in Physiotherapy".
  Potential score: 15-60 points. The higher the score, the worse the patient's situation.
  If the participant scored higher than 37.5 points at baseline, they were excluded from the study (exclusion criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Blanco-López, Physiotherapy, Principal Investigator — Universidad Católica San Antonio de Murcia (UCAM)
Locations (1):
- Clínica CEMTRO, Madrid, Madrid, Spain